CLINICAL TRIAL: NCT06041243
Title: Effects of Progressive Exercise Method Using Balance Board in Recreational Athletes With Functional Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ATADEK 2023-10/347
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Ankle Injuries
Keywords: ankle instability; game-based exercises; postural balance; physical performance; recreational athletes
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Game-based balance exercises on BoBo Home Balance Board
  Interventions: Other: Game-Based Exercises
- Control (No Intervention)

INTERVENTIONS:
Other: Game-Based Exercises — Exercises aimed to improve postural balance with four different games
  Arms: Treatment

SUMMARY:
Ankle sprains are common injuries in physically active individuals who are involved in sports such as soccer and volleyball. It is also frequently seen in sedentary individuals who are not physically active and in people who engage in recreational sports. The recurrence rate of lateral ankle sprains has been shown to be 80%. Functional Ankle Instability can be defined as recurrent ankle sprain and/or a "giving away sensation" happens after the initial sprain.

Conservative treatments are recommended to prevent recurrent injuries and to return to activity after stability, since the group that usually experiences a feeling of stability consists of young people. As a treatment, sensory and cognitive notifications and exercise applications that involve progression by increasingly challenging the individual, including reducing the support surface and changing the center of gravity, are recommended.

The Balance Board is a simple, cheap and applicable tool used to improve balance in treatment. In addition to improving balance, it reduces ankle sprains by up to 50%. The balance board can train the ankle unidirectionally or multiaxially. Unidirectional balance usually allows uniaxial movement based on a flat wood and a semicircle underneath. Multiaxial balance board systems are systems that allow multi-directional movement in all axes regardless of the position of the foot. It was reported that the performance gained as a result of the use of the multiaxial balance board was long-lasting and showed a rapid recovery in injuries. It has been concluded that balance training with a balance board restores the normal neuromuscular feedback loop by improving mechanoreceptor function, which contributes to the retraining of the sensorimotor system.

The use of game elements in treatment is defined as gamification and is a cheap and alternative method to perform various medical procedures. The increasing interest in gamification is due to lack of compliance with traditional treatment, increase in health care costs and inequitable access to health care. Musculoskeletal disorders are one of the leading causes of physical disability worldwide and gamification can be useful in various musculoskeletal rehabilitation such as tendonitis, degenerative joint disorders, neural compressions. Games are more attractive to patients and provide therapists with a wide range of alternatives for rehabilitation, making the treatment more dynamic and attractive.

The aim of our study was to investigate the effects of the exercise method on ankle stability, ankle functionality and enjoyment level of exercise in individuals with functional ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Participating recreational sports and doing at least 1.5 hours of cardiovascular or resistance training per week,
* History of one or more ankle sprains,
* Functional Ankle Instability Definition (FABIT) score >11,
* Having experienced a sprain/loss of instability in the last 6 months,
* Volunteering to attend the study.

Exclusion Criteria:

* History of an active injury in both lower extremities,
* History of surgery or fracture in both lower extremities,
* Visual, auditory and vestibular problems,
* Neurological and rheumatologic diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Star Excursion Balance Test | 4 weeks
  Straight lines are drawn on the floor in anterior, posterolateral and posteromedial directions. The individual is in the middle of these directions with the leg with instability on the floor. The other leg is asked to reach in these directions. The individual is asked to reach each of these four directions three times and the average is taken.

SECONDARY OUTCOMES:
Foot Lift Test | 4 weeks
  The individual is positioned so that the leg with instability is on the floor and the other leg is slightly flexed at the hip and knee (standing on one leg). For 30 seconds, the number of times he/she lifts the foot on the ground (e.g. lifting the toes) (including touching the opposite foot to the ground) will be tested. Three trials will be made and averaged.
Static Balance | 4 weeks
  The individual is positioned with the leg with instability on the ground and the other leg slightly flexed at the hip and knee (standing on one leg). How many seconds the individual can balance with eyes closed is measured with a stopwatch. Three trials are performed. The longest time will be evaluated. The maximum time is determined as 60 seconds.
8 Figure Jump Test | 4 weeks
  On a 5-meter-long track, the individual is asked to complete the track by jumping with the foot with instability on a path drawn in 8 shapes. It will be checked how many seconds it takes to complete the course with a stopwatch. They will be asked to make two attempts and the shortest time will be evaluated.
Side Jump Test | 4 weeks
  The individual is asked to jump 10 times with the foot with instability, 30 cm laterally and 30 cm medially. The time it takes to complete the jump is measured with a stopwatch. The individual is asked to try twice and the shortest time will be evaluated.
Short Form-12 Quality of Life Scale | 4 weeks
  It is a twelve-item questionnaire drawn from the eight subscales of the SF-36. It assesses two general health constructs: physical and mental components. All summary scores range from 0 to 100, where higher scores indicate better quality of life.
Fear-Avoidance Beliefs Questionnaire | 4 weeks
  This questionnaire can be used to assess individuals' fear-avoidance beliefs after instability. It includes an 11-question assessment. The total score ranges from 0-66. The higher the score, the higher the fear avoidance belief.
Enjoyment of Physical Activities Scale | 4 weeks
  This questionnaire aims to assess the enjoyment of the exercises in the intervention by the individuals in the study. The questionnaire consists of eight questions and each question has a score between "1-7". It is expressed as "1: strongly disagree" and "7: strongly agree". A high score indicates enjoyment of physical activity.
Global Rating of Change Scale | 4 weeks
  Individuals will be asked to mark one of the numbers "-2 -1 0 +1 +2" on a linear line to evaluate satisfaction after 4 weeks of intervention. "-2: very bad", "-1: bad", "0: same", "+1: good", "+2: very good.
Foot and Ankle Ability Measure | 4 weeks
  The Ankle Foot and Ankle Usability Measure consists of 21-questions and 2 subscales (activity of daily living (ADL) subscale and sportive activity subscale). In response to the questions, individuals are asked to mark one of the options "not difficult at all", "slightly difficult", "moderately difficult", "extremely difficult", "unable to do", "not applicable". The total score of the 21-question daily life activity section ranges from 0-84, and the total score of the 8-question sportive activity section ranges from 0-32. A higher score represents a higher functioning of each subscale. In addition, at the end of each subscale, individuals are asked to indicate their function between 0-100%. 100% indicates pre-instability function.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Mehmet Ali Aydınlar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No